CLINICAL TRIAL: NCT00692601
Title: Effect of Differing Doses of A Sweet Pepper Extract - Capsiate (A Capsaicin Analogue) - On Energy Expenditure and Blood Parameters in Humans During Exercise
Brief Title: The Acute Effects of Capsiate During Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Stuart M Phillips, Associate Professor, Department of Kinesiology, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: REB 07-410; NHPD#:130269
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Acute Exercise protocol; Crossover design; Oxygen consumption (VO2); Respiratory Exchange Ratio (RER); Adrenergic System Agonism; Capsiate Natura; Young; Male

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): acute oral ingestion of 3 mg capsiate
  Interventions: Dietary Supplement: Acute consumption of Capsiate Natura
- 2 (Experimental): acute oral ingestion of 10 mg capsiate
  Interventions: Dietary Supplement: Acute consumption of Capsiate Natura
- 3 (Placebo Comparator): acute oral ingestion of 0 mg capsiate ( same number of capsules as two other trials and identical looking placebo capsules)
  Interventions: Dietary Supplement: Acute ingestion of identical placebo capsules

INTERVENTIONS:
Dietary Supplement: Acute consumption of Capsiate Natura — 10 capsules = 3 mg total capsiate. Consumed ONCE orally as capsules 30 minutes before starting to exercise. 3 active capsules containing 1 mg capsiate each and 7 placebo capsules.
  Other Names: Brand: Capsiate Natura, Capsinoid
  Arms: 1
Dietary Supplement: Acute consumption of Capsiate Natura — 10 capsules = 10 mg total capsiate. Consumed ONCE orally as capsules 30 minutes before starting to exercise. Each capsule contains 1 mg capsiate.
  Other Names: Brand: Capsiate Natura
  Arms: 2
Dietary Supplement: Acute ingestion of identical placebo capsules — 10 mg placebo = 0 mg total capsiate. Consumed ONCE orally as capsules 30 minutes before starting to exercise. Each capsule contains 1 mg capsiate.
  Arms: 3

SUMMARY:
Capsiate is a non-pungent analogue of capsaicin, the component of hot peppers that makes them hot or spicy. Unlike capsaicin, capsiate is not spicy or hot. Ingestion of capsiate has been shown to increase resting oxygen consumption, body temperature, and the burning of fat. As such, capsiate appears to act in a manner similar to that of many other substances that energize us, increase our alertness and cause a rushing feeling by affecting a system in our body that is responsible for the release of adrenaline. The major difference, however, is that capsiate is broken down in the stomach into two components: vanilla and a fatty acid, and is not absorbed as capsiate into the blood stream at all. This implies that the way capsiate works is likely by acting on the cells in the gut (before it is broken down)rather than affecting all other cells in the body as it would do if it ended up in the blood. Therefore, the gut cells are thought to be the ones responsible for triggering the full-body adrenaline response. In any case, the use of capsiate has been shown to be effective in preventing weight gain and as such it may represent a possible therapy for treating obesity. Many obesity-related programs not involving medication advocate the use of diet and/or exercise. However, one of the biggest problems with weight loss from dieting alone is a general decrease in our body's ability to burn the food we eat as energy. This very problem is the reason for why people turn to adrenaline-releasing drugs like caffeine and ephedra. Unfortunately though, if too much is consumed, there is a high risk of bad side-effects. However, low dose caffeine/ephedra compounds (that are within specified FDA limits) have recently been reported to be effective. Moreover, these compounds are used with great frequency by people attempting to lose weight.

Given that capsiate increases body temperature, promotes the burning of body fat and has an exceptionally great side-effect profile, it looks to be a very effective supplement for use in treatment of obesity and overweight. As such, it would be important to test this supplement along with exercise. This is because consuming capsiate with exercise may enhance its effectiveness in increasing the burning of body fat. The primary purpose of this study is to examine the response of young healthy males to a 90 minute bout of moderate intensity cycling after having consumed 0 mg, 3 mg, or 10 mg of capsiate.

DETAILED DESCRIPTION:
Hypotheses

Based on the rationale and brief background above we propose the following substantive hypotheses:

1. Ingestion of capsiate 30min prior to exercise will elevate resting and exercising oxygen consumption (VO2) in a hierarchical manner: 10>3>0mg
2. Respiratory exchange ratio will be shifted toward greater lipid oxidation (i.e., toward 0.7) in a hierarchical manner: 10>3>0mg

Our secondary hypotheses are:

* A greater rise in glycerol and FFA at rest and during exercise in a hierarchical manner: 10>3>0mg
* A greater rise in catecholamine (Epinephrine and Norepinephrine) concentrations in a hierarchical manner: 10>3>0mg

Protocol We will use a double-blind repeated measures study design in which subjects will complete 3 trials - 0, 3, and 10mg - of capsiate. Based on acute effects seen in previous studies 1, 4 we anticipate that a sample size of 12 subjects (all subjects will be males to control for possible sex-based differences in substrate oxidation during exercise) would appear to be adequate to see significant effects of capsiate on oxygen consumption and substrate oxidation. Randomization will be done on a counterbalanced and blocked basis with 3 conditions and 6 possible order combinations and with 12 subjects, each subject will be randomized in a counterbalanced manner so that 2 subjects complete each trial order.: ABC, ACB, BCA, BAC, CAB, CBA, order of treatment and assignment will be performed at random and under complete control of the McMaster University Pharmacy. The chief pharmacist - Dr. Gita Sobhi - will give the code for each treatment to the PI only after completion of the data analysis. We will use a cycling protocol at an intensity of 55% of each subject's individual peak VO2 for 90 minutes. Workload to determine 55% of peak VO2 will be according to the algorithm detailed by Latin et al. 17 This exercise intensity is adequate to elevate lipolysis (i.e., glycerol and FFA), catecholamines, and show a substantial shift in RER toward lipid oxidation with increasing exercise duration. The PI has experience with this protocol and has measured substrate oxidation previously using the same or very similar protocols. 18-20 Moreover, this type of exercise intensity represents an intensity that elicits an exercising RER in or around 0.9 and thus where there is a good blend (65:35 carbohydrate:lipid) of fuels being oxidized, but is also an intensity close to what has been referred to as 'fatmax', which is defined as the intensity of exercise at which the maximal rate of lipid oxidation occurs. 16, 21-23 Thus, in terms of selecting an exercise intensity that will reveal the impact of capsiate on both energy expenditure and substrate oxidation we believe that this intensity is an optimal one. We will collect breath (breath-by-breath and ensemble averaged into 30s bins) and blood samples for 30min into recovery to assess to what degree excess post-exercise oxygen consumption is elevated and whether this is accompanied by significant fat oxidation and elevated plasma catecholamines.

We will use recreationally active subjects (peak VO2 > 40 ml/kg/min) so that we're assured they will be able to complete the protocol. Subjects will be screened using a standard health questionnaire (see attached consent form) and a maximal exercise test. Subjects will be healthy non-smokers between the ages of 18-30 and will be recruited from the local McMaster University campus or surrounding community. Exercise trials will take place in the overnight fasted state (last meal at 2000h) after having consumed a standardized diet on the day prior to the exercise trial. Having subjects in the fasted state does not present a risk or barrier to the subjects completing the trial as based on past experience with this protocol. It is emphasized that being in the fasted state is also the easiest state in which to interpret the data from the standpoint of substrate oxidation. The pre-trial day diet will consist of energy estimated for each subject based on the Harris-Benedict equation 24 with an activity factor of 40%. The diet will be 50:30:20 in terms of percent energy from carbohydrate:fat:protein. Subjects will consume the same diet on the days prior to each exercise trial to control for pre-study calorie and carbohydrate/fat intake, which could affect substrate oxidation. Subjects will refrain from consumption of alcohol and caffeine on the day of the trial. Trials will take place at least 5d (but no more than 7d) apart and will commence at a time between ~7-10am and will proceed according to the schematic timeline shown in figure 1. The testing time for subjects will remain consistent throughout the study. We also believe that it is prudent for subjects to consume a fixed and constant volume of water (1000ml) during all trials to prevent dehydration and to allow subjects to complete the ride in safe manner.

All data will be analyzed using a repeated measures two-way analysis of variance with time as a within factor and dose as a between factor. Significant ANOVA effects will be further scrutinized using Tukey's test as a post-hoc procedure. Where significant correlation of one variable with another exists an analysis of covariance may also be performed. Significance will be accepted at P<0.05.

Analysis VO2 and RER for energy expenditure and substrate use - standard equations using revised non-protein RER as described by Jeukendrup and Wallis. 26 HR - using Polar™ monitoring and on-line collection via the AEI metabolic cart BP - using Finapres™ blood pressure monitoring. Blood glucose, glycerol, lactate - fluorometric methods as detailed in Passoneau and Lowry 27 and as performed previously by the PI. 18, 20, 28 Free fatty acids - colorimetric micro-assay method from WAKO diagnostics (http://www.wakodiagnostics.com/r_nefa.html) Catecholamines - using reverse phase HPLC and electrochemical detection as described previously. 18, 20

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Recreationally active
* Non-smokers
* Age 18-30 years
* Favourable (low risk) answers on Standard Health Questionnaire (part of approved consent form)
* Peak VO2 of > 40 ml/kg/min
* Recruited from the local McMaster University campus or surrounding community.

Exclusion Criteria:

* Women
* Smokers
* Contraindicated health conditions which would render someone "clinically" unhealthy i.e. diabetes, liver, kidney abnormalities, etc.
* Possible allergies to the study products (Capsiate or Placebo)
* The use of foods, other natural health products or pharmaceuticals that may interact with the study products
* The use of natural health products that alter the outcome measures of the trial

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Respiratory Exchange Ratio (RER) for substrate use | breath by breath analysis of oxygen uptake and carbon dioxide release (recorded as the average oxygen uptake and carbon dioxide relsease every 30 seconds)

SECONDARY OUTCOMES:
Heart Rate | measured 8 times over 180 minutes
Blood Pressure monitoring | measured 8 times over 180 minutes
Blood biomarkers (blood glucose, glycerol, lactate, Free fatty acids [FFA]) | measured 6 times over 180 minutes
Plasma Catecholamines (Epinephrine, norepinephrine) | measured 6 times over 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D., Principal Investigator — Department of Kinesiology, McMaster University; Andrea R Josse, M.Sc., Study Director — Department of Kinesiology, McMaster University; Nicholas A Burd, M.Sc., Study Director — Department of Kinesiology, McMaster University; Yoshiyuki Fujishima, D.Phil., Study Chair — Ajinomoto USA, INC.
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Masuda Y, Haramizu S, Oki K, Ohnuki K, Watanabe T, Yazawa S, Kawada T, Hashizume S, Fushiki T. Upregulation of uncoupling proteins by oral administration of capsiate, a nonpungent capsaicin analog. J Appl Physiol (1985). 2003 Dec;95(6):2408-15. doi: 10.1152/japplphysiol.00828.2002. Epub 2003 Sep 5. PMID 12959953
- [Background] Ohnuki K, Haramizu S, Oki K, Watanabe T, Yazawa S, Fushiki T. Administration of capsiate, a non-pungent capsaicin analog, promotes energy metabolism and suppresses body fat accumulation in mice. Biosci Biotechnol Biochem. 2001 Dec;65(12):2735-40. doi: 10.1271/bbb.65.2735. PMID 11826971
- [Background] Ohnluki K, Haramizu S, Watanabe T, Yazawa S, Fushiki T. CH-19 sweet, nonpungent cultivar of red pepper, increased body temperature in mice with vanilloid receptors stimulation by capsiate. J Nutr Sci Vitaminol (Tokyo). 2001 Aug;47(4):295-8. doi: 10.3177/jnsv.47.295. PMID 11767210
- [Background] Ohnuki K, Niwa S, Maeda S, Inoue N, Yazawa S, Fushiki T. CH-19 sweet, a non-pungent cultivar of red pepper, increased body temperature and oxygen consumption in humans. Biosci Biotechnol Biochem. 2001 Sep;65(9):2033-6. doi: 10.1271/bbb.65.2033. PMID 11676017